CLINICAL TRIAL: NCT00831792
Title: An Observational Study of Continuous TKI258, in Castration-Resistant Prostate Cancer Patients Evaluating Markers of FGF Signaling in Bone Marrow Plasma
Brief Title: TKI258 in Castrate Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0510; NCI-2011-01106 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-01-27; First posted 2009-01-29 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Advanced Prostate Cancer; Castrate Resistant Prostate Cancer; Prostate Specific Antigen; PSA; Castration-Resistant Prostate Cancer Patients; TK1258; CHIR-258
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TK1258 (Experimental): 4 capsules (100 mg/capsules) of TKI 258 by mouth once daily (total of 400 mg of TKI258 per day). Following an initial 4-week cycle at a starting dose of 400 mg 5 days- on and 2 days off, TKI258 may be escalated to 500 mg/day 5 days-on/2 days off if no significant Grade3/4 AEs or laboratory abnormalities are observed.
  Interventions: Drug: TK1258

INTERVENTIONS:
Drug: TK1258 — 4 capsules (100 mg/capsules) of TKI 258 by mouth once daily (total of 400 mg of TKI258 per day).
  Other Names: CHIR-258

SUMMARY:
The goal of this clinical research study is to learn if a decrease in the levels of prostate specific antigen (PSA) may be linked with the status of prostate cancer that has spread to the bones. Researchers also want to learn how changes in your blood PSA level might affect the rebuilding of healthy bones while you are being treated with TKI258 for prostate cancer.

DETAILED DESCRIPTION:
The Study Drug:

TKI258 is designed to perform several anti-tumor functions, including cutting off the blood supply to tumors. Researchers think this may help slow or stop the growth of prostate cancer.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take 4 capsules of TKI258 1 time each day for 5 days in a row followed by 2 days of rest (Days 1-5, 8-12, 15-19, and 22-26 of each 28-day study "cycle"). You should take the TKI258 capsules with about 8 ounces of water and at least 1 hour before a meal (breakfast) or at least 2 hours following a meal (breakfast). If you want, you may take the drug with a meal that has fewer than 500 calories and 20 grams of fat.

Study Visits:

Every 28 days makes up 1 study "cycle."

On Day 1 of Cycle 1 and all cycles after that, the following tests and procedures will be performed:

* Your complete medical history will be recorded.
* You will be asked about any drugs or treatments you may be receiving.
* You will be asked about any side effects you may have experienced.
* You will have a physical exam, including measurement of your vital signs and weight.
* Your performance status will be evaluated.
* Blood (about 2 tablespoons) will be collected for routine tests. This blood will also be tested to measure your PSA.
* You will have a triplicate ECG (3 ECGs in a row) before you take the study drug. You will also have 1 ECG about 6 hours after you take the study drug.

On Day 12 (+/- 3 days) of Cycles 1 and 2, and day 26 of Cycle 1 (+/- 3 days) blood (about 1 tablespoon) will be collected for routine tests. Part of the Cycle 2 blood draw will be used to measure the amount of TKI258 in your system. Note that the Day 26 of Cycle 1 visit could end up being scheduled on the same day as the Day 1 of Cycle 2 visit described above.

On Day 1 of Cycle 2 and every odd numbered Cycle after this (Cycles 3, 5, 7and so on), the following tests and procedures will be performed:

* Blood (about 2 teaspoons) will be collected for routine tests.
* Urine will be collected to test for markers relating to your bone.

At the end of every cycle (about Day 26), you will have an ECG.

Every 3 Cycles (about every 12 weeks), the following tests and procedures will be performed:

* Blood (about 1 teaspoon) will be drawn to measure your levels of heart enzymes
* You will have an echocardiogram or MUGA scan like the one you had at the screening visit to check your heart function.

About 7-10 weeks after your first dose of study drug, you will have another bone marrow biopsy and aspiration performed to check the status of the disease and for biomarker testing.

CT and/or bone scans will be performed every 8 weeks for the first 6 months and every 3 months after that to check the status of the disease.

Length of Study:

You may remain on study for as long as you are benefiting. You will be taken off study if intolerable side effects occur or if the disease gets worse.

End-of-Study Visit:

Within 4 weeks after your last dose of the study drug, you will return to the clinic for an end-of-study visit. The following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs, and weight.
* Your performance status will be evaluated.
* You will be asked about any drugs or treatments you may be receiving.
* You will be asked about any side effects you have experienced since you last visit.
* Blood (about 3 tablespoons) and urine will be collected for routine tests. This blood will also be tested to measure certain hormones, heart enzymes, and PSA.
* You will have a chest x-ray, bone scan, and either a computed tomography (CT) or magnetic resonance imaging (MRI) scan of your abdomen and pelvis to check the status of the disease.
* You will have an ECG and either an echocardiogram or a MUGA scan.
* You will have a bone marrow biopsy and aspiration performed to check the status of the disease and for biomarker testing.

Long-Term Follow-up:

Once you are no longer on this study, the research staff will check up on you about every 3 months. This update will consist of a phone call, an e-mail, or a review of your medical and/or other records. You will not have any extra tests, procedures, or study visits. If contacted by phone, the call would only last about 5 minutes.

This is an investigational study. TKI258 is not FDA approved or commercially available. It is being used in this study for research purposes only.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven adenocarcinoma of the prostate with evidence for skeletal metastases on bone scan and/or CT scan.
2. Eastern Cooperative Oncology Group (ECOG) performance status </= 2. (Karnofsky Performance Status >/= 50%)
3. Serum testosterone levels </= 50ng/ml
4. Ongoing gonadal androgen deprivation therapy with luteinizing hormone-releasing hormone (LHRH) analogues or orchiectomy. Patients, who have not had an orchiectomy, must be maintained on standard dosing of LHRH analogue therapy at appropriate frequency for the duration of the study.
5. Progression of disease despite androgen ablation (either documented osseous or soft tissue metastatic disease progression or by PSA criteria progression). a)Definition of Progressive disease by PSA evidence: a PSA level of at least 5 ng/ml which has risen on at least 2 successive occasions, at least 2 weeks apart. The participant will need a baseline test and a test to show that the PSA has increased.
6. Discontinue diethylstilbestrol (DES) for >/= 4 weeks and antiandrogens >/= 6 weeks prior to study drug.
7. Discontinue any steroids prescribed to specifically treat prostate cancer (for e.g as a secondary hormonal manipulation or for cord compression) >/= 4 weeks prior to study drug. Steroids chronically prescribed for a non-cancer-related illness (e.g. asthma or COPD) that is well controlled with medical management are permissible to an equivalent of < 10 mg Prednisone daily.
8. Antiandrogen Withdrawal: Patients who are receiving an antiandrogen as part of primary androgen ablation must demonstrate disease progression following discontinuation of antiandrogen. Disease progression after antiandrogen withdrawal is defined as 2 consecutive rising PSA values, obtained at least 2 weeks apart, or documented osseous or soft tissue progression.
9. For patients receiving flutamide, at least one of the PSA values must be obtained 4 weeks or more after flutamide discontinuation.
10. For patients receiving bicalutamide or nilutamide, at least one of the PSA values must be obtained 6 weeks or more after antiandrogen discontinuation
11. Laboratory Requirements: 1) Adequate adrenal function (absence of symptoms or electrolyte imbalances that indicate adrenal insufficiency); 2) White blood cell count (WBC) count >/= 3,000/microl; 3) Absolute Neutrophil Count (ANC) >/= 1,500/microl; 4) Hemoglobin >/= 8.0 g/dL independent of transfusion; 5) Platelet count >/= 75,000/microL; 6) Serum albumin >/= 3.0 g/dL; 7) Serum creatinine < 1.5 x ULN or a calculated creatinine clearance > 60 mL/min (as calculated by Cockcroft-Gault method) 8) Serum potassium >/= 3.5 mmol/L
12. No evidence of chronic or acute DIC (Disseminated Intravascular Coagulation) or bleeding tendency and no angina at rest.
13. Patient must be willing and able to comply with protocol requirements. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must also have signed an authorization for the release of their protected health information.

Exclusion Criteria:

1. Histologic variants other than adenocarcinoma in the primary tumor
2. Abnormal liver functions consisting of any of the following: a) Serum bilirubin >/= 1.5 * upper limit of normal (ULN) b) AST and ALT > 2.5 * ULN
3. Therapy with other hormonal therapy, including any dose of Ketoconazole, finasteride (Proscar), dutasteride (Avodart) any herbal product known to decrease PSA levels (eg, Saw Palmetto and PC-SPES) within 4 weeks of study drug.
4. Requirement for corticosteroids greater than the equivalent of 7.5 mg of prednisone daily.
5. Therapy with samarium or strontium within 8 weeks prior to first dose of study drug.
6. Active infection or concomitant illness that is not controlled with medical management.
7. Prior radiation therapy completed < 4 weeks or single fraction of palliative radiotherapy within 14 days prior to first dose of study drug.
8. Any currently active second malignancy, other than non-melanoma skin cancer. Patients are not considered to have a currently active malignancy, if they have completed therapy and are considered by their physician to be at least less than 30% risk of relapse over next 3 months.
9. Active psychiatric illnesses/social situations that would limit compliance with protocol requirements.
10. Active or uncontrolled autoimmune disease that may require corticosteroid therapy during study
11. Severely compromised immunological state, including being positive for the human immunodeficiency virus (HIV)
12. Acute or chronic hepatitis B or C
13. Chemotherapy and other investigational therapies (targeted or immunotherapy) will require a 4-week washout period before treatment initiation
14. Initiation of bisphosphonate therapy within 4 weeks prior to first dose of study drug. Patients on stable doses of bisphosphonates that show subsequent tumor progression may continue on this medication; however, patients are not allowed to initiate bisphosphonate therapy during the study.
15. Impaired cardiac function or clinically significant cardiac diseases, including any of the following: a.) History or presence of serious uncontrolled ventricular arrhythmias or presence of atrial fibrillation; b.) Clinically significant resting bradycardia (< 50 beats per minute); c.) Left ventricular ejection fraction (LVEF) assessed by 2-D echocardiogram (ECHO) < 50% or lower limit of normal (whichever is higher) or multiple gated acquisition scan (MUGA) < 45% or lower limit of normal (whichever is higher);
16. (# 13 Conti'd) Any of the following within 6 months prior to study entry: myocardial infarction (MI), severe/unstable angina, Coronary Artery Bypass Graft (CABG), Congestive Heart Failure (CHF), Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA), Pulmonary Embolism (PE); e.) Uncontrolled hypertension defined by an SBP>150 and/or a DBP>100 mm Hg with or without anti-hypertensive medication; f.) Previous pericarditis; clinically significant pleural effusion in the previous 12 months or current ascites requiring 2 or more interventions per month.
17. History of pituitary or adrenal dysfunction
18. History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug.
19. Prior therapy with TKI258
20. Any acute toxicities due to prior chemotherapy and/or radiotherapy that have not resolved to a National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (version 3.0) grade of </= 1. Chemotherapy induced alopecia and grade 2 neuropathy is allowed.
21. Condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study.
22. Men whose partner is a woman of child-bearing potential, (i.e. biologically able to conceive), and who is not employing two forms of highly effective contraception. Highly effective contraception (e.g. male condom with spermicide, diaphragm with spermicide, intra-uterine device) must be used by both sexes during the study and must be continued for 8 weeks after the end of study treatment. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Women of child-bearing potential is defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (e.g., who has had menses any time in the preceding 12 consecutive months).

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-04-07 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Corn, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Castration-Resistant Prostate Cancer patients were enrolled between 2010-2013
Groups:
- Eligible Patients: All patients enrolled and treated with TKI 258
Period: Overall Study
Arm/Group | Eligible Patients
Started | 46
Completed | 40
Not Completed | 6
Not completed — Not Eligible | 3
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Groups:
- All Patients Enrolled and Treated With TKI 258: Patients with castrate-resistant prostate cancer
Arm/Group | All Patients Enrolled and Treated With TKI 258
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 33
Age, Continuous [Mean (Full Range); unit: years] | 69 [57 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 41
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Improvement, Disease Progression or Stable Disease
Description: Three consecutive PSA elevations above nadir or baseline are required for progression. Each increment in PSA should be a minimum of 1 ng/ml and at least 2 weeks apart or will not count. The time of PSA progression will be taken as the time of the first of these PSA elevations that represents an increment by at least 25% above the nadir or baseline. Given that increments in PSA do not always represent treatment failure, particularly when novel agents with uncertain effects on PSA levels are being evaluated, clinical and radiological correlation is recommended at the discretion of the treating physician. In patients with PSA progression alone without clinical or radiological evidence of disease progression, continued therapy on study is at the discretion of the treating physician in consultation with the principal investigator.
Time Frame: From the time of enrollment until 30 days beyond the date of the last study drug administration
Population: Patients completed at least 1 cycle of therapy
Measure: Count of Participants; unit: Participants
Groups:
- APatients on Observational Study of TKI258: Patients with histologically confirmed adenocarcinoma of the prostate with bone metastases
Arm/Group | APatients on Observational Study of TKI258
Number analyzed (Participants) | 23
Participants
  Bone scan/soft tissue mets improvements at 8 wks | 6
  Disease progression | 4
  experienced stable disease at 8 weeks | 13

ADVERSE EVENTS:
Time Frame: From the time of enrollment until 30 days beyond the date of the last study drug administration
Arm/Group | All Patients Enrolled and Treated With TKI 258
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 2/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients Enrolled and Treated With TKI 258 (N=40)
Muscle weakness, generalized or specific area (not due to neuropathy): Extremity - lower (Musculoskeletal and connective tissue disorders) | 1
Infection with unknown ANC--Select: Urinary tract NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils--Select: Skin (cellulitis) (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients Enrolled and Treated With TKI 258 (N=40)
Alkaline phosphatase (Metabolism and nutrition disorders) | 23
Allergy/Immunology-Other (Specify) (Immune system disorders) | 1
Alopecia (Endocrine disorders) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Hepatobiliary disorders) | 10
Amylase (Metabolism and nutrition disorders) | 4
Anemia (Metabolism and nutrition disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 22
AST, SGOT (serum glutamic oxaloacetic transaminase) (Hepatobiliary disorders) | 15
Ataxia (incoordination) (Nervous system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Atrophy, skin (Skin and subcutaneous tissue disorders) | 1
Autoimmune reaction (Immune system disorders) | 1
Back pain (Vascular disorders) | 4
Bilirubin (hyperbilirubinemia) (Hepatobiliary disorders) | 2
Bladder spasms (Renal and urinary disorders) | 2
Bone pain (Vascular disorders) | 2
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Vascular disorders) | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 9
Chest wall pain (Vascular disorders) | 2
Cholesterol, serum-high (hypercholestremia) (Metabolism and nutrition disorders) | 1
Confusion (Nervous system disorders) | 2
Constipation (Gastrointestinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Creatinine (Metabolism and nutrition disorders) | 7
Cystitis noninfective (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dehydration (Gastrointestinal disorders) | 6
Depression (Psychiatric disorders) | 1
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 31
DIC (disseminated intravascular coagulation) (Vascular disorders) | 1
Dizziness (Nervous system disorders) | 2
Dry mouth/salivary gland (xerostomia) (General disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4
Dysesthesia (Nervous system disorders) | 2
Dysgeusia (Gastrointestinal disorders) | 3
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 11
Edema limbs (Vascular disorders) | 2
Edema trunk (Vascular disorders) | 1
Edema: limb (Vascular disorders) | 12
Edema: trunk/genital (Vascular disorders) | 1
Fatigue (asthenia, lethargy, malaise) (Metabolism and nutrition disorders) | 39
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10^9 per liter) (Infections and infestations) | 3
fibrinogen (Blood and lymphatic system disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastrointestinal-Other (Specity) (General disorders) | 1
GGT (gamma-Glutamyl transpeptidase) (Hepatobiliary disorders) | 8
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3
Headache (Nervous system disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Hemoglobin (Blood and lymphatic system disorders) | 25
Hemoglobinuria (Renal and urinary disorders) | 1
Hemorrhage, GU--Select (Urinary NOS) (Renal and urinary disorders) | 1
Hot flashes (Endocrine disorders) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 21
Hypertension (Adult) (Cardiac disorders) | 3
Hypoalbuminemia (Hepatobiliary disorders) | 13
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Hypotension (Cardiac disorders) | 4
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1
Incontinence (Renal and urinary disorders) | 4
Infection with normal ANC or Grade 1 or 2 neutrophils--Select (Urinary tract NOS) (Infections and infestations) | 1
Infection (clinically or microbiologically) (Infections and infestations) | 1 — with Grade 3 or 4 neutrophils (ANC <1.0 x 10^9 per liter
Infection without neutropenia (Infections and infestations) | 1
Infection-Other (Specify) (Infections and infestations) | 3
INR (International Normalized Ratio of prothrombin time) (Metabolism and nutrition disorders) | 1
Insomnia (Nervous system disorders) | 6
Leukocytes (Total WBC) (Blood and lymphatic system disorders) | 8
Lipase (Metabolism and nutrition disorders) | 2
Localized edema (Vascular disorders) | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 2
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 7
Mood alteration-depression (Psychiatric disorders) | 1
Mood alteration--Select (Psychiatric disorders) | 1
Mood alteration--Select (Depression) (Psychiatric disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam) (Oral Cavity) (Gastrointestinal disorders) | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy) (Extremity - lower) (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness, generalized or specific area (not due to neuropathy) (Whole body/generalized) (Musculoskeletal and connective tissue disorders) | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 26
Neurology-Other (Specify) (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 12
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 5
Non-cardiac chest pain (Cardiac disorders) | 1
Pain (Vascular disorders) | 3
Pain in extremity (Vascular disorders) | 1
Pain-Other (Specify) (Vascular disorders) | 19
Pain--Select (Abdomen NOS) (Vascular disorders) | 5
Pain--Select (Back) (Vascular disorders) | 17
Pain--Select (Bone) (Vascular disorders) | 8
Pain--Select (Buttock) (Vascular disorders) | 1
Pain--Select (Cardiac/heart) (Vascular disorders) | 1
Pain--Select (Chest wall) (Vascular disorders) | 1
Pain--Select (Dental/teeth/peridontal) (Vascular disorders) | 1
Pain--Select (Extremity-limb) (Vascular disorders) | 6
Pain--Select (Head/headache) (Vascular disorders) | 3
Pain--Select (Joint) (Vascular disorders) | 4
Pain--Select (Liver) (Vascular disorders) | 1
Pain--Select (Pain NOS) (Vascular disorders) | 3
Pain--Select (Pelvis) (Vascular disorders) | 6
Pain--Select (Rectum) (Vascular disorders) | 1
Pain--Select (Scalp) (Vascular disorders) | 1
Pain--Select (Throat/pharynx/larynx) (Vascular disorders) | 1
Pancreatic endocrine: glucose intolerance (Endocrine disorders) | 1
Paresthesia (Nervous system disorders) | 1
Pelvic pain (Vascular disorders) | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2
Platelets (Blood and lymphatic system disorders) | 12
Pleural effusion (non-malignant) (Cardiac disorders) | 2
Potassium serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 4
Proteinuria (Metabolism and nutrition disorders) | 5
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 3
Pulmonary/Upper Respiratory-Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 13
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Rigors, chills (Infections and infestations) | 2
Salivary gland changes/saliva (Gastrointestinal disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 1
Supraventricular and nodal arrhythmia--Select (Atrial fibrillation) (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia--Select (Atrial flutter) (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia--Select (Sinus tachycardia) (Cardiac disorders) | 2
Syncope (fainting) (Nervous system disorders) | 2
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 4
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 3
Tooth infection (General disorders) | 1
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 9
Urinary tract infection (Infections and infestations) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Urinary tract pain (Renal and urinary disorders) | 1
Urine color change (Renal and urinary disorders) | 2
Vision-blurred vision (Eye disorders) | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 14
Watery eye (epiphora, tearing) (Eye disorders) | 4
Weight loss (Metabolism and nutrition disorders) | 6
White blood cell decreased (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-05-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT00831792/Prot_SAP_000.pdf